CLINICAL TRIAL: NCT03448211
Title: A Phase I Open-Label, Dose-Escalation Study of Para-toluenesulfonamide Injection (PTS) Administered Intratumorally and Locally to Patients With Solid Tumors
Brief Title: A Study of PTS for Patients With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development strategy reasons
Sponsor: PTS International Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: US-01
Record Dates: First submitted 2018-02-06; First posted 2018-02-28 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — 4-toluenesulfonamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Para-toluenesulfonamide Injection (PTS) (Experimental): Investigational product
  Interventions: Drug: Para-toluenesulfonamide Injection (PTS)

INTERVENTIONS:
Drug: Para-toluenesulfonamide Injection (PTS) — Intratumoral injection
  Other Names: PTS

SUMMARY:
The primary objective of this study is to determine the MTD of PTS following local and intratumoral injections over a treatment course of two 5-day cycles to patients with palpable advanced solid malignancies who have failed standard treatment.

DETAILED DESCRIPTION:
The study will be an open, uncontrolled, single-center, phase I study to assess the safety and tolerability of local intra-tumoral injection 2.0ml (660mg), 4.0ml (1220mg), 6.0ml (1880mg) and 8.0ml (2440mg) PTS in female breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are diagnosed as unsuitable for surgical operations or refuse to do so.
* Subject's performance status is classified as Grade 0 to Grade 3. Estimated survival time should be longer than 6 months of time.
* Physical examinations show no serious functional disorders of the heart, liver, kidneys, or blood.
* Subjects were treated with radio or chemotherapy previously. A minimum of 2 to 3 months recovery time is required before treating with this investigational drug.
* Subject is diagnosed as intratracheal lesions with metastasized pulmonary cancer not suitable for surgery, or refuses to be operated.
* Subject should show lobular atelectasis with either complete or incomplete obstruction of the bronchi.
* Physical examinations should show no functional disorders of the heart, liver, kidneys, central nervous system, and blood.
* Subject performance status to be classified from Grade 0 to Grade 3, who can tolerate the fiberoptic bronchoscopy treatments.
* In-patient is preferred. When subject is in satisfactory conditions, the out Cpatient can also be enrolled in this trial.
* Two to three months recovery time is required for the subject has just received radio or chemotherapy.
* Emergency request, subjects with serious lobular atelectasis and almost complete obstruction of the bronchi.
* With the aid of a tracheal intubation and the help of the respirator, PTS may be intraumorally injected into the obstructed lesion via fiberoptic bronchoscopy outside of the tube, alongside of the intubation.

Exclusion Criteria:

* Pregnant women and children will not be used as test subjects.
* Subjects with serious functional disorders of the heart, liver, kidneys, or blood will be excluded.
* Subjects who do not want to participate in the trial will not be used as test subjects.
* Subject does not agree to participate.
* Subject performance status is Grade 4, and the one who does not want to tolerate the discomfort of the PTS treatments via fiberoptic bronchscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose | 4 weeks post-treatment
  Maximum tolerable dose

CONTACTS AND LOCATIONS:
Overall Officials: Nan-Shan Zhong, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States